CLINICAL TRIAL: NCT05031429
Title: Time Limited Eating in New-Onset Type 1 Diabetes: Feasibility, Acceptability, and Effect on β-cell Function
Brief Title: Time Limited Eating in Type 1 Diabetes
Acronym: TLET1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, jennifer raymond, Chief of the Division of Endocrinology, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-21-00269
Record Dates: First submitted 2021-08-01; First posted 2021-09-01 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Time Limited Eating; β-cell
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard Care (No Intervention): * includes a minimum 12-hour feeding window for 7 days per week
  * no caloric restriction will be used
  * will wear a continuous glucose monitor
- Intervention - Time Limited Eating (Experimental): * includes an 8-hour feed/16-hour fast for 7 days per week
  * will be instructed to consume all of their calories in the afternoon/evening period
  * can consume non-caloric beverages (water, tea, coffee) during the fasting period
  * will wear a continuous glucose monitor
  * no caloric restriction will be used
  Interventions: Other: Time Limited Eating

INTERVENTIONS:
Other: Time Limited Eating — Includes an 8-hour feed/16-hour fast for 7 days per week, with consumption of all of calories in the afternoon/evening. Can consume non-caloric beverages (water, tea, coffee) during the fasting period. No caloric restriction will be used.
  Arms: Intervention - Time Limited Eating

SUMMARY:
This study is a randomized-control pilot study that aims to evaluate Time Limited Eating (TLE) in the pediatric T1D population, implemented within the first six months after diagnosis. This period is characterized by residual β-cell function, during which TLE may have the ability to preserve and improve β-cell activity, indicated by increased C-peptide production. The investigators aim to assess the feasibility, acceptability, and safety of TLE in the pediatric T1D population, as well as to investigate the impact of TLE on β-cell function, insulin sensitivity, and glycemic control.

DETAILED DESCRIPTION:
This will be a two-armed study with an intervention and control group. Feasibility and acceptability will be assessed by using questionnaires. Safety will be indicated by hypoglycemia occurrence. β-cell function and insulin sensitivity will be evaluated using mixed meal tolerance test with C-peptide and glucose levels. Glycemic control will be indicated by continuous glucose monitor (CGM). Block randomization will be utilized to ensure the groups are balanced in terms of BMI. The study period will be 9 weeks in duration, including a week-long run-in period and an 8-week intervention period. There will be two in-person study visits at week 0 and week 9. Anthropometrics including weight, height, and pubertal status will be evaluated at these times.

Group 1- Standard Care (control)

* includes a minimum 12-hour feeding window for 7 days per week
* no caloric restriction will be used
* will wear a continuous glucose monitor

Group 2 - TLE (intervention)

* includes an 8-hour feed/16-hour fast for 7 days per week
* will be instructed to consume all of their calories in the afternoon/evening period
* can consume non-caloric beverages (water, tea, coffee) during the fasting period
* will wear a continuous glucose monitor
* no caloric restriction will be used

ELIGIBILITY:
Inclusion Criteria:

* includes age of 12-25 years
* T1D diagnosed within 6 months
* at least one positive pancreatic antibody including glutamic acid decarboxylase (GAD) antibody, islet tyrosine phosphatase 2 (IA2) antibody, or insulin antibody
* can be on either insulin injections or insulin pump
* can be of any BMI status
* can speak any language

Exclusion Criteria:

* negative pancreatic antibodies
* unwillingness to wear a CGM

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility of intervention, as indicated by the "Intervention Satisfaction Survey" | At end of study (at 9 weeks)
  Likert scale "Agree strongly" is 1, "Agree" is 2, "Neutral" is 3, "Disagree" is 4, and "Disagree strongly" is 5. Lower scores indicate more satisfaction, higher scores indicate low satisfaction.
Change in β-cell function at 9 weeks, as indicated by mixed meal tolerance test with C-peptide levels | Baseline and 9 weeks
  C-peptide and glucose levels will be performed at baseline and 60-, 90-, and 120-minutes post-meal. Baseline plasma C-peptide concentration divided by the baseline plasma glucose concentration will be calculated as a pragmatic marker of β-cell function. The area under the stimulated C-peptide curve will then be calculated, which will be the primary outcome examined.
Change in glycemic control at 9 weeks, as indicated by continuous glucose monitoring (percent time in range), and HbA1c | Up to 9 weeks; HbA1c: Baseline and 9 weeks
  Continuous glucose monitors will be worn for duration of the study, glycemic control will be evaluated using percent time in range. HbA1c will reflect glycemic control over time.
Safety, as indicated by hypoglycemia | Up to 9 weeks
  Hypoglycemia will be defined as blood sugar < 70 mg/dL on continuous glucose monitor. Frequency and severity of hypoglycemia will be used to assess safety of intervention.

SECONDARY OUTCOMES:
Dietary patterns, as indicated by the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) | Baseline, 9 weeks
  24-hour dietary recall, ~30 minutes to complete.
Quality of life, as indicated by Pediatric Quality of Life Inventory (PedsQL), Diabetes Module | Baseline and 9 weeks
  Likert scale "Never" is 0, "Almost Never" is 1, "Sometimes" is 2, "Often" is 3, and "Almost Always" is 4
Stress level, as indicated by Perceived Stress Scale | Baseline and 9 weeks
  Likert scale "Never" is 0, "Almost Never" is 1, "Sometimes" is 2, "Fairly Often" is 3, and "Very Often" is 4
Binge Eating, as indicated by Binge Eating Disorder Screener | Baseline and 9 weeks
  Likert scale "Never or rarely" is 0, "Sometimes" is 1, "Often" is 2, "Always" is 3. Additionally, two yes or no questions.
Anxiety, as indicated by Neuro-QOL-Anxiety-Short Form | Baseline and 9 weeks
  Likert scale "Never" is 1, "Rarely" is 2, "Sometimes" is 3, "Often" is 4, "Always" is 5
Impact on activities of daily living, as indicated by Munich Chronotype Questionnaire (MCTQ) | Baseline and 9 weeks
  Assessment of sleep schedule, school schedule, time spent outdoors. Multiple choice and open-ended questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabel K, Varady KA. Feasibility of Time-Restricted Eating. Obesity (Silver Spring). 2020 May;28(5):860. doi: 10.1002/oby.22785. No abstract available. PMID 32320147
- [Background] Gabel K, Hoddy KK, Varady KA. Safety of 8-h time restricted feeding in adults with obesity. Appl Physiol Nutr Metab. 2019 Jan;44(1):107-109. doi: 10.1139/apnm-2018-0389. Epub 2018 Sep 14. PMID 30216730
- [Background] Cienfuegos S, Gabel K, Kalam F, Ezpeleta M, Wiseman E, Pavlou V, Lin S, Oliveira ML, Varady KA. Effects of 4- and 6-h Time-Restricted Feeding on Weight and Cardiometabolic Health: A Randomized Controlled Trial in Adults with Obesity. Cell Metab. 2020 Sep 1;32(3):366-378.e3. doi: 10.1016/j.cmet.2020.06.018. Epub 2020 Jul 15. PMID 32673591
- [Background] Wilkinson MJ, Manoogian ENC, Zadourian A, Lo H, Fakhouri S, Shoghi A, Wang X, Fleischer JG, Navlakha S, Panda S, Taub PR. Ten-Hour Time-Restricted Eating Reduces Weight, Blood Pressure, and Atherogenic Lipids in Patients with Metabolic Syndrome. Cell Metab. 2020 Jan 7;31(1):92-104.e5. doi: 10.1016/j.cmet.2019.11.004. Epub 2019 Dec 5. PMID 31813824
- [Background] Taylor R. Type 2 diabetes: etiology and reversibility. Diabetes Care. 2013 Apr;36(4):1047-55. doi: 10.2337/dc12-1805. No abstract available. PMID 23520370
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Hutchison AT, Regmi P, Manoogian ENC, Fleischer JG, Wittert GA, Panda S, Heilbronn LK. Time-Restricted Feeding Improves Glucose Tolerance in Men at Risk for Type 2 Diabetes: A Randomized Crossover Trial. Obesity (Silver Spring). 2019 May;27(5):724-732. doi: 10.1002/oby.22449. Epub 2019 Apr 19. PMID 31002478
- [Background] Chow LS, Manoogian ENC, Alvear A, Fleischer JG, Thor H, Dietsche K, Wang Q, Hodges JS, Esch N, Malaeb S, Harindhanavudhi T, Nair KS, Panda S, Mashek DG. Time-Restricted Eating Effects on Body Composition and Metabolic Measures in Humans who are Overweight: A Feasibility Study. Obesity (Silver Spring). 2020 May;28(5):860-869. doi: 10.1002/oby.22756. Epub 2020 Apr 9. PMID 32270927
- [Background] Jamshed H, Beyl RA, Della Manna DL, Yang ES, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves 24-Hour Glucose Levels and Affects Markers of the Circadian Clock, Aging, and Autophagy in Humans. Nutrients. 2019 May 30;11(6):1234. doi: 10.3390/nu11061234. PMID 31151228
- [Background] Center for Disease and Control Prevention. Incidence of newly diagnosed diabetes. https://www.cdc.gov/diabetes/data/statistics-report/newly-diagnosed-diabetes.html. 2020; Accessed April 25, 2021.
- [Background] Bingley PJ, Wherrett DK, Shultz A, Rafkin LE, Atkinson MA, Greenbaum CJ. Type 1 Diabetes TrialNet: A Multifaceted Approach to Bringing Disease-Modifying Therapy to Clinical Use in Type 1 Diabetes. Diabetes Care. 2018 Apr;41(4):653-661. doi: 10.2337/dc17-0806. PMID 29559451
- [Background] Lennerz BS, Barton A, Bernstein RK, Dikeman RD, Diulus C, Hallberg S, Rhodes ET, Ebbeling CB, Westman EC, Yancy WS Jr, Ludwig DS. Management of Type 1 Diabetes With a Very Low-Carbohydrate Diet. Pediatrics. 2018 Jun;141(6):e20173349. doi: 10.1542/peds.2017-3349. Epub 2018 May 7. PMID 29735574
- [Background] de Souza Bosco Paiva C, Lima MHM. Introducing a very low carbohydrate diet for a child with type 1 diabetes. Br J Nurs. 2019 Aug 8;28(15):1015-1019. doi: 10.12968/bjon.2019.28.15.1015. PMID 31393762
- [Background] Calabrese CM, Valentini A, Calabrese G. Gut Microbiota and Type 1 Diabetes Mellitus: The Effect of Mediterranean Diet. Front Nutr. 2021 Jan 13;7:612773. doi: 10.3389/fnut.2020.612773. eCollection 2020. PMID 33521039
- [Background] Vidmar AP, Goran MI, Naguib M, Fink C, Wee CP, Hegedus E, Lopez K, Gonzalez J, Raymond JK. Time limited eating in adolescents with obesity (time LEAd): Study protocol. Contemp Clin Trials. 2020 Aug;95:106082. doi: 10.1016/j.cct.2020.106082. Epub 2020 Jul 16. PMID 32682994
- [Background] Liu H, Javaheri A, Godar RJ, Murphy J, Ma X, Rohatgi N, Mahadevan J, Hyrc K, Saftig P, Marshall C, McDaniel ML, Remedi MS, Razani B, Urano F, Diwan A. Intermittent fasting preserves beta-cell mass in obesity-induced diabetes via the autophagy-lysosome pathway. Autophagy. 2017;13(11):1952-1968. doi: 10.1080/15548627.2017.1368596. Epub 2017 Nov 25. PMID 28853981
- [Background] Brandhorst S, Choi IY, Wei M, Cheng CW, Sedrakyan S, Navarrete G, Dubeau L, Yap LP, Park R, Vinciguerra M, Di Biase S, Mirzaei H, Mirisola MG, Childress P, Ji L, Groshen S, Penna F, Odetti P, Perin L, Conti PS, Ikeno Y, Kennedy BK, Cohen P, Morgan TE, Dorff TB, Longo VD. A Periodic Diet that Mimics Fasting Promotes Multi-System Regeneration, Enhanced Cognitive Performance, and Healthspan. Cell Metab. 2015 Jul 7;22(1):86-99. doi: 10.1016/j.cmet.2015.05.012. Epub 2015 Jun 18. PMID 26094889
- [Background] Cheng CW, Villani V, Buono R, Wei M, Kumar S, Yilmaz OH, Cohen P, Sneddon JB, Perin L, Longo VD. Fasting-Mimicking Diet Promotes Ngn3-Driven beta-Cell Regeneration to Reverse Diabetes. Cell. 2017 Feb 23;168(5):775-788.e12. doi: 10.1016/j.cell.2017.01.040. PMID 28235195
- [Background] Foster NC, Beck RW, Miller KM, Clements MA, Rickels MR, DiMeglio LA, Maahs DM, Tamborlane WV, Bergenstal R, Smith E, Olson BA, Garg SK. State of Type 1 Diabetes Management and Outcomes from the T1D Exchange in 2016-2018. Diabetes Technol Ther. 2019 Feb;21(2):66-72. doi: 10.1089/dia.2018.0384. Epub 2019 Jan 18. PMID 30657336
- [Background] DuBose SN, Hermann JM, Tamborlane WV, Beck RW, Dost A, DiMeglio LA, Schwab KO, Holl RW, Hofer SE, Maahs DM; Type 1 Diabetes Exchange Clinic Network and Diabetes Prospective Follow-up Registry. Obesity in Youth with Type 1 Diabetes in Germany, Austria, and the United States. J Pediatr. 2015 Sep;167(3):627-32.e1-4. doi: 10.1016/j.jpeds.2015.05.046. Epub 2015 Jul 8. PMID 26164381
- [Background] Tommerdahl KL, Baumgartner K, Schafer M, Bjornstad P, Melena I, Hegemann S, Baumgartner AD, Pyle L, Cree-Green M, Truong U, Browne L, Regensteiner JG, Reusch JEB, Nadeau KJ. Impact of Obesity on Measures of Cardiovascular and Kidney Health in Youth With Type 1 Diabetes as Compared With Youth With Type 2 Diabetes. Diabetes Care. 2021 Mar;44(3):795-803. doi: 10.2337/dc20-1879. Epub 2021 Jan 5. PMID 33402367
- [Background] Bjornstad P, Snell-Bergeon JK, Rewers M, Jalal D, Chonchol MB, Johnson RJ, Maahs DM. Early diabetic nephropathy: a complication of reduced insulin sensitivity in type 1 diabetes. Diabetes Care. 2013 Nov;36(11):3678-83. doi: 10.2337/dc13-0631. Epub 2013 Sep 11. PMID 24026551
- [Background] Bjornstad P, Schafer M, Truong U, Cree-Green M, Pyle L, Baumgartner A, Garcia Reyes Y, Maniatis A, Nayak S, Wadwa RP, Browne LP, Reusch JEB, Nadeau KJ. Metformin Improves Insulin Sensitivity and Vascular Health in Youth With Type 1 Diabetes Mellitus. Circulation. 2018 Dec 18;138(25):2895-2907. doi: 10.1161/CIRCULATIONAHA.118.035525. PMID 30566007
- [Background] Ruan Y, Willemsen RH, Wilinska ME, Tauschmann M, Dunger DB, Hovorka R. Mixed-meal tolerance test to assess residual beta-cell secretion: Beyond the area-under-curve of plasma C-peptide concentration. Pediatr Diabetes. 2019 May;20(3):282-285. doi: 10.1111/pedi.12816. Epub 2019 Feb 19. PMID 30652426
- [Background] Shim WS, Kim SK, Kim HJ, Kang ES, Ahn CW, Lim SK, Lee HC, Cha BS. Decrement of postprandial insulin secretion determines the progressive nature of type-2 diabetes. Eur J Endocrinol. 2006 Oct;155(4):615-22. doi: 10.1530/eje.1.02249. PMID 16990662
- [Background] Paglialunga S, Guerrero A, Roessig JM, Rubin P, Dehn CA. Adding to the spectrum of insulin sensitive populations for mixed meal tolerance test glucose reliability assessment. J Diabetes Metab Disord. 2016 Dec 7;15:57. doi: 10.1186/s40200-016-0279-x. eCollection 2016. PMID 27981043
- [Background] Shankar SS, Vella A, Raymond RH, Staten MA, Calle RA, Bergman RN, Cao C, Chen D, Cobelli C, Dalla Man C, Deeg M, Dong JQ, Lee DS, Polidori D, Robertson RP, Ruetten H, Stefanovski D, Vassileva MT, Weir GC, Fryburg DA; Foundation for the National Institutes of Health beta-Cell Project Team. Standardized Mixed-Meal Tolerance and Arginine Stimulation Tests Provide Reproducible and Complementary Measures of beta-Cell Function: Results From the Foundation for the National Institutes of Health Biomarkers Consortium Investigative Series. Diabetes Care. 2016 Sep;39(9):1602-13. doi: 10.2337/dc15-0931. Epub 2016 Jul 12. PMID 27407117
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Bergman RN, Phillips LS, Cobelli C. Physiologic evaluation of factors controlling glucose tolerance in man: measurement of insulin sensitivity and beta-cell glucose sensitivity from the response to intravenous glucose. J Clin Invest. 1981 Dec;68(6):1456-67. doi: 10.1172/jci110398. PMID 7033284
- [Background] Shah VN, DuBose SN, Li Z, Beck RW, Peters AL, Weinstock RS, Kruger D, Tansey M, Sparling D, Woerner S, Vendrame F, Bergenstal R, Tamborlane WV, Watson SE, Sherr J. Continuous Glucose Monitoring Profiles in Healthy Nondiabetic Participants: A Multicenter Prospective Study. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4356-4364. doi: 10.1210/jc.2018-02763. Erratum In: J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1775-e1776. doi: 10.1210/clinem/dgab837. PMID 31127824
- [Background] Harnack L. Nutrition Data System for Research (NDSR). In: Gellman M.D., Turner J.R. (eds) Encyclopedia of Behavioral Medicine. Springer. 2013.
- [Background] Raper N, Perloff B, Ingwerson L, Steinfeldt L, Anand J. An overview of USDA's Dietary Intake Data System. Journal of Food Composition and Analysis. 2004;17(3-4):545-555.
- [Background] Hood KK, Beavers DP, Yi-Frazier J, Bell R, Dabelea D, Mckeown RE, Lawrence JM. Psychosocial burden and glycemic control during the first 6 years of diabetes: results from the SEARCH for Diabetes in Youth study. J Adolesc Health. 2014 Oct;55(4):498-504. doi: 10.1016/j.jadohealth.2014.03.011. Epub 2014 May 10. PMID 24815959
- [Background] Ivezaj V, White MA, Grilo CM. Examining binge-eating disorder and food addiction in adults with overweight and obesity. Obesity (Silver Spring). 2016 Oct;24(10):2064-9. doi: 10.1002/oby.21607. Epub 2016 Aug 25. PMID 27558207
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Vidmar AP, Goran MI, Raymond JK. Time-Limited Eating in Pediatric Patients with Obesity: A Case Series. J Food Sci Nutr Res. 2019;2(3):236-244. doi: 10.26502/jfsnr.2642-11000022. Epub 2019 Sep 20. PMID 32455345